CLINICAL TRIAL: NCT01803022
Title: Prescription and Utilization of Low Molecular Weight Heparin in Usual Medical Practice for the Curative Treatment of Venous Thromboembolism in Patients With Cancer
Status: Completed | Type: Observational
Sponsor: LEO Pharma (Industry)
Responsible Party: Sponsor
Other Study IDs: Tropique
Record Dates: First submitted 2013-02-26; First posted 2013-03-04 (Estimated); Last update posted 2018-02-05 (Actual); Status verified 2018-02

CONDITIONS: Venous Thromboembolism
Keywords: Venous Thromboembolism; Cancer; Low Molecular Weight Heparin
MeSH Terms: conditions — Venous Thromboembolism; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Low Molecular Weight Heparin

SUMMARY:
The study purpose is to document the prescription and the use of Low Molecular Weight Heparin in usual medical practice in patients with cancer and established Venous Thromboembolism. This study also aims at gathering epidemiological data on the Low Molecular Weight Heparin therapy of Venous Thromboembolism in patients with cancer.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must provide informed consent
* Men or women aged 18 years or more
* Ongoing cancer disease recent diagnosis of veinous thromboembolism treatment with Low Molecular Weight Heparin before entry into the study

Exclusion Criteria:

- Contraindication to the use of Low Molecular Weight Heparin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men or women aged 18 years or more with on-going cancer and recent diagnosis of Venous Thromboembolism, treated with Low Molecular Weight Heparin before entry into the study
Sampling Method: Probability Sample
Enrollment: 419 (Actual)
Dates: Start 2012-11; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Prescription conditions and use of Low Molecular Weight Heparin in the French usual practice for the treatment of symptomatic Venous Thromboembolism in patients with cancer at up to 6 months | up to 6 months

SECONDARY OUTCOMES:
To evaluate the consistency of the Low Molecular Weight Heparin use with French national recommendations on the treatment of Venous Thromboembolism in patients with cancer. | up to 6 months
To evaluate Venous Thromboembolism recurrences, bleeding, thrombocytopenia and deaths during Low Molecular Weight Heparin treatment | up to 6 months
To describe clinical factors associated with treatment duration with Low Molecular Weight Heparin and those associated with the occurrence of Venous Thromboembolism in patients with cancer | up to 6 months
To evaluate the anticoagulant treatment perception and satisfaction by patients with cancer disease with a validated questionnaire | up to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Dominique Farge Bancel, Pr, Principal Investigator — Groupe Francophone Thrombose et Cancer
Locations (1):
- Hopital Saint Louis, Paris, France

IPD SHARING:
Plan to Share IPD: No